CLINICAL TRIAL: NCT02492191
Title: RAPP- Systematic E-assessment of Postoperative Recovery in Patients Undergoing Day Surgery
Acronym: RAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Ulrica Nilsson, Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-4765
Record Dates: First submitted 2015-07-05; First posted 2015-07-08 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Postoperative Complications
Keywords: Smart Phones; Ambulatory Care; Outcome and Process Assessment
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RAPP, e- assessed follow-up (Active Comparator): A mobile application (app) is installed on each patient's own smartphone. The app includes the Swedish web version of the QoR (SwQoR). After a patient is discharged from the day-surgery department, the patients in the intervention group will answer the RAPP daily for 14 days. His or her smartphone will initiate the postoperative recovery measurements daily through a "push" function. Each question will appear separately on the mobile phone screen and will disappear from the screen immediately after a response is given. The app also contains a question asking if the patient wants to be contacted by a nurse, which they will answer with a YES or NO. If YES, a nurse at the day surgery department will contact the patient and offer further information and assistance. The number of contacts and the reasons for contact requests will be documented.
  Interventions: Device: Smartphone app Recovery Assessment by Phone Points (RAPP)
- Control (No Intervention): The control group will receive standard care; i.e., no follow-up

INTERVENTIONS:
Device: Smartphone app Recovery Assessment by Phone Points (RAPP) — An e-assessed follow-up of day surgery patients postoperative recovery measured via smartphone app
  Arms: RAPP, e- assessed follow-up

SUMMARY:
Introduction Day surgery is a well-established practice in many European countries, but only limited information is available regarding postoperative recovery at home though there is a current lack of a standard procedure regarding postoperative follow-up. Furthermore, there is also a need for improvement of modern technology in assessing patient related outcomes such as native software applications. This article describes the RAPP study protocol, a mixed-methods study to evaluate if a systematic e-assessment follow-up in patients undergoing day surgery is cost effective and improves postoperative recovery, health and quality of life.

Methods and analysis This study is a mixed-methods study design that includes a multicenter, two-group, parallel, single-blind randomized controlled trial (RCT) and qualitative interview studies. One thousand patients >17 years of age who are undergoing day surgery will be randomly assigned to either e-assessed postoperative recovery follow-up daily in 14 days measured via smartphone app including the Swedish web-version of Quality of Recovery (SwQoR) or to standard care (i.e. no follow up). The primary aim is cost effectiveness. Secondary aims are improvements on postoperative recovery, health-related quality of life (QoL) and overall health; (b) to determine whether differences in health literacy have a substantial and distinct effect on postoperative recovery, health, and QoL; and (c) to describe day-care patient and staff experiences with a systematic e-assessment follow-up after day surgery.The primary will be measured at 2 weeks postoperatively and secondary outcomes b) at 1 and 2 weeks and c) at 1 and 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Understand the Swedish language in speech and writing, have an Android or iPhone OS smartphone, and give their informed consent to participate

Exclusion Criteria:

* Undergoing abortion, if their journal entries indicate alcohol and/or drug abuse or memory impairment, if they are participating in another clinical trial or suffering from visual impairment. .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1046 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Cost effectiveness | 14 days postoperatively
  The analysis of cost effectiveness will consider the costs associated with the follow-up, gained QALYs from SF-6D. The SF-6D provides a means for using the SF-36 by estimating a preference-based single-index measure for health from these data using general population values. This analysis will be complemented with information regarding the individuals' willingness to pay for the follow-up, number of healthcare contacts, and duration and degree of sick leave.

SECONDARY OUTCOMES:
Postoperative recovery | 7 and 14 days postoperatively
  All participants will evaluate their postoperative recovery using the SwQoR. Participants in the intervention group will answer by using the smartphone app, and those in the control group will use a conventional paper-based questionnaire.
Quality of Life (QoL) | Preoperatively(baseline) and 14 days postoperatively
  QoL will be assessed with the SF-36
Overall health | Preoperatively(baseline) and 14 days postoperatively
  Overall health will be measured by the EQ visual analog scale (EQ-VAS). This scale consists of a vertically graduated scale with endpoints (anchors) of 0 indicating worst imaginable health state and 100 indicating best imaginable health state
Health literacy | 14 days postoperatively
  To measure health literacy (i.e., the equality perspective), we will use the Japanese Communicative and Critical Health Literacy scale (C&CHL scale), which includes items covering the major aspects of communicative and critical health literacy. The C&CHL scale has been translated into Swedish and demonstrated to be understandable, stable over time, and equivalent to the Japanese C&CHL scale in terms of language and content
Patient experience of the intervention | 1 month postopertively
  Following the RCT, inductive qualitative research will be conducted to explore the perceptions, views, experiences, and expectations of the participants from the intervention group. Data will be collected based on 20 semistructured interviews. A purposeful sampling will be conducted. Patients who wished to be contacted by a nurse via the RAPP during the intervention period will be selected, with variation regarding age and gender. The aim of this study is to explore the participants' experience of postoperative recovery and how using the RAPP for postoperative follow-up influenced this recovery. Further questions will be asked regarding the participants' experience of being contacted by a nurse; in addition, descriptions and eventual expectations about the help that was received will also be solicited. All interviews will be recorded and transcribed verbatim.
Staff experience of the implementation | 4 months postoperatively
  As part of this RCT, we will also describe the staffs' experience of using a systematic postoperative follow-up tool and their willingness to pay for the follow-up service. We plan to make the data from the patients' daily postoperative recovery measurements available to the staff at the day-surgery departments and to record the experiences and opinions of the clinicians. The study design will be qualitative and will use focus-group interviews. One to two focus-group interviews with 5-8 participants each will be conducted at each hospital, depending on the size of the day-surgery department. Staff from the day-surgery department (nurses, surgeons, and anesthesiologists) will be asked to participate in the interviews. All interviews will be recorded and transcribed verbatim.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrica Nilsson, Prof, Principal Investigator — Faculty of Medicine and Health, Örebro University, Sweden
Locations (1):
- Örebro university hospital, Day surgery department, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson U, Jaensson M, Dahlberg K, Odencrants S, Gronlund A, Hagberg L, Eriksson M. RAPP, a systematic e-assessment of postoperative recovery in patients undergoing day surgery: study protocol for a mixed-methods study design including a multicentre, two-group, parallel, single-blind randomised controlled trial and qualitative interview studies. BMJ Open. 2016 Jan 13;6(1):e009901. doi: 10.1136/bmjopen-2015-009901. PMID 26769788
- [Background] Jaensson M, Dahlberg K, Eriksson M, Gronlund A, Nilsson U. The Development of the Recovery Assessments by Phone Points (RAPP): A Mobile Phone App for Postoperative Recovery Monitoring and Assessment. JMIR Mhealth Uhealth. 2015 Sep 11;3(3):e86. doi: 10.2196/mhealth.4649. PMID 26362403
- [Derived] Nilsson U, Dahlberg K, Jaensson M. Swedish Web Version of the Quality of Recovery Scale Adapted for Patients Undergoing Local Anesthesia and Peripheral Nerve Blockade (SwQoR-LA): Prospective Psychometric Evaluation Study. JMIR Perioper Med. 2021 Jan 15;4(1):e23090. doi: 10.2196/23090. PMID 33448932
- [Derived] Jaensson M, Dahlberg K, Nilsson U. Sex Similarities in Postoperative Recovery and Health Care Contacts Within 14 Days With mHealth Follow-Up: Secondary Analysis of a Randomized Controlled Trial. JMIR Perioper Med. 2018 Mar 26;1(1):e2. doi: 10.2196/periop.9874. PMID 33401367
- [Derived] Halleberg Nyman M, Nilsson U, Dahlberg K, Jaensson M. Association Between Functional Health Literacy and Postoperative Recovery, Health Care Contacts, and Health-Related Quality of Life Among Patients Undergoing Day Surgery: Secondary Analysis of a Randomized Clinical Trial. JAMA Surg. 2018 Aug 1;153(8):738-745. doi: 10.1001/jamasurg.2018.0672. PMID 29710226
- [Derived] Dahlberg K, Philipsson A, Hagberg L, Jaensson M, Halleberg-Nyman M, Nilsson U. Cost-effectiveness of a systematic e-assessed follow-up of postoperative recovery after day surgery: a multicentre randomized trial. Br J Anaesth. 2017 Nov 1;119(5):1039-1046. doi: 10.1093/bja/aex332. PMID 29077819
- [Derived] Jaensson M, Dahlberg K, Eriksson M, Nilsson U. Evaluation of postoperative recovery in day surgery patients using a mobile phone application: a multicentre randomized trial. Br J Anaesth. 2017 Nov 1;119(5):1030-1038. doi: 10.1093/bja/aex331. PMID 29077818